CLINICAL TRIAL: NCT00170469
Title: A Phase II, Dose Ranging Multi-Centre, Single Blind, Parallel-Group, Controlled Study of the Safety, Tolerability and Immunogenicity of Recombinant (rPA Based) Anthrax Vaccine Compared With Anthrax Vaccine Adsorbed in a Healthy Population
Brief Title: Safety, Tolerability and Immunogenicity of Recombinant Anthrax Vaccine Compared With Anthrax Vaccine Adsorbed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmAthene UK Limited (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05-0002; PA-8645-02
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Bacillus Anthracis (Anthrax)
Keywords: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Low dose rPA vaccine
  Interventions: Biological: rPA vaccine containing alhydrogel
- 2 (Experimental): High dose rPA vaccine
  Interventions: Biological: rPA vaccine containing alhydrogel
- 3 (Active Comparator): Active vaccine control
  Interventions: Biological: AVA

INTERVENTIONS:
Biological: AVA
  Arms: 3
Biological: rPA vaccine containing alhydrogel
  Arms: 1; 2

SUMMARY:
This is a dose ranging study comparing different vaccine schedules of rPA vaccine, for Anthrax, to the licensed dose of AVA, another Anthrax vaccine. Safety and the capability to induce an immune response will be evaluated.

DETAILED DESCRIPTION:
Anthrax is a zoonotic disease, occurring in wild and domestic mammals, caused by the spore-forming bacterium Bacillus anthracis (B. anthracis). Anthrax occurs in humans when they are exposed to infected animals, tissue from infected animals or when they are directly exposed to B. anthracis or its spores. Depending on the route of infection, anthrax disease can occur in three forms: cutaneous, gastrointestinal, and inhalation. In the United States of America (USA), the annual incidence of human anthrax has declined from approximately 130 cases annually in the early 1900s to no cases during 1999 to 2000. However, in the USA, shortly after September 11th, 2001, there were 22 cases (18 confirmed) of inhaled and cutaneous anthrax infection that were related to contaminated mail. The development of a new anthrax vaccine is necessary because the current AVA vaccine requires the growth of B. anthracis in its manufacturing process and has a complex administration regimen of six administrators of vaccine in 18 months. As protective antigen (PA) is a central virulence factor in anthrax pathogenesis and a major immunogen in the current vaccine, a recombinant, acellular, protective antigen-based anthrax vaccine, could offer an improved manufacturing process and a simpler dosing schedule. Furthermore, the vaccine could offer improved protection against inhaled B. anthracis, and could, when used in conjunction with antibiotics, form part of the management of anthrax exposed individuals. This is a dose ranging study comparing different primary vaccine schedules of rPA Anthrax vaccine to the licensed dose of Anthrax Vaccine Adsorbed. The study is designed to measure the immune response, and to evaluate the safety and tolerability of different doses of rPA Anthrax Vaccine. After subjects have given informed consent, they will undergo physical exams, medical history screening, pregnancy tests, ECG, HIV, Hepatitis B & C tests, safety blood tests, and urine drug and alcohol screen. Subjects will be asked to complete a diary card to record any symptoms they may experience. The subjects that receive AVA will be offered the opportunity to complete the licensed course of vaccination which would involve AVA vaccinations at 6, 12 and 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females.
2. Aged between 18-55 years (inclusive).
3. A body mass index (BMI) of 18-35.
4. Signed informed consent, which includes information about the potential risks and effects of rPA and AVA.
5. A medical history without major organ pathology (e.g. cardiac, immunological, psychiatric, endocrine or neurological disorders, cancer or other wasting diseases - (adequately treated actinic keratosis, or basal cell carcinoma [BCC], or carcinoma in situ [CIS] of the cervix are permitted).
6. A female may be enrolled if one of the following criteria applies:

   Either If of child-bearing capacity then: A female is not pregnant or breast feeding AND is routinely using adequate injectable or transdermal (administered at the recommended frequency) or oral contraception (at a stable dose for at least three months prior to the first dose of vaccine) and will continue to do so during the study, augmenting this contraceptive measure with a barrier method OR is sexually abstinent OR is monogamous and has a partner who has had a vasectomy (>1 month previously) OR is using a commonly recognized copper and hormone implanted intrauterine device (IUD) such as TCu-380A, TCu-220C, MLCu-375, Nova-T, or LNG-20. In addition, the subject must have a negative blood pregnancy test prior to enrolment into the study and negative urine pregnancy test pre-dose.

   Or A female is post menopausal (defined as a female with no menstrual cycle for at least 24 months and of menopausal age (>45 years) Or A female with no menstrual cycle for between 12 and 24 months and of menopausal age (>45 years) who has a negative blood pregnancy test prior to enrolment into the study and a negative urine pregnancy test pre-dose.

   Or A female has been surgically sterilized (confirmed by review of medical record).

   Or A female has had a total hysterectomy at least 3 months prior to the start of the study (confirmed by review of medical record).
7. A male may be enrolled if willing to use barrier methods of contraception and whose partner is using an acceptable form of contraception for 3 months post each dose.

Exclusion Criteria:

1. Presence of any clinically significant medical condition as determined by the Investigator.
2. Medically significant hypersensitivity or idiosyncratic reaction related to any medical product including vaccines.
3. History or evidence of drug abuse 1 year prior to enrollment.
4. Participation in a clinical study of an investigational vaccine within 3 months prior to the start of the study or an investigational drug product within 30 days prior to the start of the study.
5. Use of any prescription or non-prescription medication within 7 days prior to the first dosing with the exception of over-the-counter (OTC) antihistamine, non-steroidal anti-inflammatory drugs (NSAID), acetaminophen, OTC decongestants or oral/injectable/transdermal contraceptives. Any medication taken within 7 days of the first dosing will be recorded.
6. History or suspicion of inability to co-operate adequately.
7. Donation of blood or blood products for a period of 4 weeks prior to participation in the study.
8. Immunodeficiency or clinically active autoimmune disease.
9. Positive urine alcohol and drug screen for drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, and barbiturates).
10. Positive test for human immunodeficiency virus (HIV), and/or hepatitis B and/or hepatitis C.
11. Vaccination(s) with a live vaccine in the previous 4 weeks or killed / inactivated vaccines in the previous 3 weeks.
12. Blood or plasma transfusions, or pooled gamma-globulin in the previous 3 months and need for blood or plasma transfusions during this study.
13. Received anthrax vaccine or anthrax immune globulin or been otherwise exposed to B. anthracis.
14. Clinically relevant abnormal findings on routine physical examination.
15. Clinically significant out-of-range laboratory tests at screening including: urinalysis, serum creatine, lactate dehydrogenase (LDH), potassium, glucose, liver function tests (LFT); absolute neutrophil count, platelet count, white blood cell count, electrolytes, clotting and blood hemoglobin.
16. Twelve-lead ECG recording with clinically relevant signs of pathology and conduction disturbances as judged by the investigator.
17. Presence of tattoos that cover or partially cover the injection sites on the upper arm.
18. Known sensitivity to Latex.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2005-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety of rPA vaccine

SECONDARY OUTCOMES:
Immunogenicity of rPA vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Currie, MD, Principal Investigator — Accelovance
Locations (16):
- United States (16):
  - Greater Huntsville Family Practice, PC, Huntsville, Alabama
  - Discovery Alliance, Inc., Mobile, Alabama
  - Accelovance, San Diego, California
  - Accelovance, Washington D.C., District of Columbia
  - Florida Medical Research Institute, Gainesville, Florida
  - Accelovance, Melbourne, Florida
  - Miami Research Associates, South Miami, Florida
  - Accelovance, Orland Park, Illinois
  - Accelovance, South Bend, Indiana
  - Accelovance, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - McKenzie Medical Center, McKenzie, Tennessee
  - PharamTex Research, Inc., Amarillo, Texas
  - Accelovance, Houston, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Carilion Medical Associates, Galax, Virginia